CLINICAL TRIAL: NCT05938166
Title: The Effects of Using Augmented Reality (AR) System to Train Foreign Care on Salivary Biomarker and Oral Function of the Elderly People
Brief Title: The Effects of Using Augmented Reality (AR) System to Train Foreign Care Workers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUHIRB-SV(II)-20230019
Record Dates: First submitted 2023-07-03; First posted 2023-07-10 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Oral Dryness and Saliva Altered; Oral Manifestations; Swallowing Disorder
Keywords: AR (augmented reality); Oral Care Behavior; Saliva Biomarker
MeSH Terms: conditions — Xerostomia; Oral Manifestations; Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- experimental group (EG-A) (Experimental): Behavioral: The experimental of A group received a 40-minute AR tooth-cleaning skills session and a 50-minute video-based oral hygiene education course.
  Interventions: Device: oral care augmented reality (AR); Other: video-based oral hygiene education course
- experimental group (EG-B) (Experimental): The experimental of B group received a 50-minute video-based oral hygiene education course.
  Interventions: Other: video-based oral hygiene education course
- Control Group (No Intervention): The CG only receive only a booklet of traditional classroom oral health education

INTERVENTIONS:
Device: oral care augmented reality (AR) — Augmented reality (AR) is an extension of perceptible reality, whereby additional information, such as texts or virtual objects, can be displayed in the user's field of vision.The oral care augmented reality (AR) simulation training can train foreign care workers by switching languages (Indonesian) and therefore reduce language-related learning barriers.
  Arms: experimental group (EG-A)
Other: video-based oral hygiene education course — 50-minute video-based oral hygiene education course
  Arms: experimental group (EG-A); experimental group (EG-B)

SUMMARY:
The aim of this study was to evaluate the effect of augmented reality (AR) system training intervention of foreign care workers on the salivary biomarker and oral function of older people.

This randomized controlled trial included experimental group: AR group (EG-A) Video group (EG-B) and control group(CG), respectively. The EG-A will receive augmented reality (AR) system training intervention with AR tooth-cleaning skills session course add video-based oral hygiene education course . The EG-B receive video-based oral hygiene education course and The CG only receive only a leaflet.

DETAILED DESCRIPTION:
A randomized experimental design was used. Female foreign care workers whose aged 21 to 65 years and by cared older peoples whose aged 65 to 75 years were recruited through community-based site of long-term care service in Kaohsiung city. Each group was expected for 12 care workers and by cared older peoples who each group. G*Power (version 3.1.9.4) was used for power analysis.

All foreign care workers whose participants will underwent questionnaire examination at baseline and at 1-month, 3-month, 6-month follow-ups. The information of foreign care workers regarding oral care cognition, attitude, self-efficacy, and oral care behavior intention will be collected by a self-report questionnaire before and after intervention.

Each by cared older peoples will be evaluation oral hygiene and function by oral hygienist, and will completed the questionnaire at baseline and at 1-month, 3-month and 6-month follow-up. Older people by cared will assess plaque control record (PCR), tongue coating index (TCI), repetitive saliva swallowing test (RSST), oral diadochokinetic (DDK), oral moisture degree (OMD),masticatory efficiency (MoE) and salivary biomarker at baseline (Time 1), three months (Time 2) and six months (Time 3) follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 1. The Indonesian caregivers who are employed in Kaohsiung City are aged between 21 and 65 and have simple Chinese communication skills.
* 2. The elderly people being cared for is over 65 years old.

Exclusion Criteria:

* 1. Elderly people who are unable to cooperate with instructions.
* 2. Elderly people with facial impairment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tongue Coating Index(TCI) | Change from Baseline TCI at 1-month after intervention
  The tongue-coating status of 9 areas of tongue surfaces was recorded using the tongue coating index, as follows:
  Score 0: Tongue coating not visible.
  Score 1: Tongue coating thin, papillae of tongue visible.
  Score 2: Tongue coating very thick, papillae of tongue not visible.
  Range= 0 to 18 Score
Tongue Coating Index(TCI) | Change from Baseline TCI at 3-month after intervention
  The tongue-coating status of 9 areas of tongue surfaces was recorded using the tongue coating index, as follows:
  Score 0: Tongue coating not visible.
  Score 1: Tongue coating thin, papillae of tongue visible.
  Score 2: Tongue coating very thick, papillae of tongue not visible.
  Range= 0 to 18 Score
Tongue Coating Index(TCI) | Change from Baseline TCI at 6-month after intervention
  The tongue-coating status of 9 areas of tongue surfaces was recorded using the tongue coating index, as follows:
  Score 0: Tongue coating not visible.
  Score 1: Tongue coating thin, papillae of tongue visible.
  Score 2: Tongue coating very thick, papillae of tongue not visible.
  Range= 0 to 18 Score
Oral Dryness Status | Change from Baseline Oral Dryness Status at 1-month after intervention
  The oral dryness status of saliva flow rate was recorded using the saxon test(Chew gauze sponge for 2 mins), as follows:
  Normal: 2.75 g/2min.
  Oral dryness: 2 g/2min.
Oral Dryness Status | Change from Baseline Oral Dryness Status at 3-month after intervention
  The oral dryness status of saliva flow rate was recorded using the saxon test(Chew gauze sponge for 2 mins), as follows:
  Normal: 2.75 g/2min.
  Oral dryness: 2 g/2min.
Oral Dryness Status | Change from Baseline Oral Dryness Status at 6-month after intervention
  The oral dryness status of saliva flow rate was recorded using the saxon test(Chew gauze sponge for 2 mins), as follows:
  Normal: 2.75 g/2min.
  Oral dryness: 2 g/2min.
Lip-Tongue Motor Function | Change from Baseline lip-tongue motor function Status at 1-month after intervention
  The lip-tongue motor function status of count-by-time was recorded using the Oral diadochokinesis rate (lip-tongue function (Pa/ Ta /Ka) in syllables or times per 15 seconds), as follows:
  Pa:times/ per 15 seconds
  Ta:times /per 15 seconds
  Ka:times /per 15 seconds
Lip-Tongue Motor Function | Change from Baseline lip-tongue motor function Status at 3-month after intervention
  The lip-tongue motor function status of count-by-time was recorded using the Oral diadochokinesis rate (lip-tongue function (Pa/ Ta /Ka) in syllables or times per 15 seconds), as follows:
  Pa:times/ per 15 seconds
  Ta:times /per 15 seconds
  Ka:times /per 15 seconds
Lip-Tongue Motor Function | Change from Baseline lip-tongue motor function Status at 6-month after intervention
  The lip-tongue motor function status of count-by-time was recorded using the Oral diadochokinesis rate (lip-tongue function (Pa/ Ta /Ka) in syllables or times per 15 seconds), as follows:
  Pa:times/ per 15 seconds
  Ta:times /per 15 seconds
  Ka:times /per 15 seconds
Maximum tongue pressure (MTP) | Change from Baseline Maximum tongue pressure status at 1-month after intervention
  The tongue pressure of 3 times pressure average was recorded using the Maximum tongue pressure test, as follows:
  1. First times / Maximum Kpa value.
  2. Second times / Maximum Kpa value.
  3. Third times / Maximum Kpa value.
  Average of maximum tongue pressure in 3 times.
Maximum tongue pressure (MTP) | Change from Baseline Maximum tongue pressure status at 2-month after intervention
  The tongue pressure of 3 times pressure average was recorded using the Maximum tongue pressure test, as follows:
  1. First times / Maximum Kpa value.
  2. Second times / Maximum Kpa value.
  3. Third times / Maximum Kpa value.
  Average of maximum tongue pressure in 3 times.
Maximum tongue pressure (MTP) | Change from Baseline Maximum tongue pressure status at 3-month after intervention
  The tongue pressure of 3 times pressure average was recorded using the Maximum tongue pressure test, as follows:
  1. First times / Maximum Kpa value.
  2. Second times / Maximum Kpa value.
  3. Third times / Maximum Kpa value.
  Average of maximum tongue pressure in 3 times.
Masticatory Function | Change from Baseline Change from Baseline Maximum tongue pressure status at 1-month after intervention status at 3-month after intervention
  The mixing ability was assessed using color-changeable chewing gum (Masticatory Performance Evaluating Gum XYLITOL, Lotte, Tokyo, Japan) , as follows:
  To chew as usual on the gum 120 seconds. The chewing rhythm was kept constant at once per second.color scale consisting of five intermediate colors .
  1. light green: very poor chewing ability.
  2. light yellow: poor chewing ability.
  3. light pink: no good chewing ability.
  4. pink: good chewing ability.
  5. red: very good chewing ability.
Masticatory Function | Change from Baseline Change from Baseline Maximum tongue pressure status at 3-month after intervention status at 3-month after intervention
  The mixing ability was assessed using color-changeable chewing gum (Masticatory Performance Evaluating Gum XYLITOL, Lotte, Tokyo, Japan) , as follows:
  To chew as usual on the gum 120 seconds. The chewing rhythm was kept constant at once per second.color scale consisting of five intermediate colors .
  1. light green: very poor chewing ability.
  2. light yellow: poor chewing ability.
  3. light pink: no good chewing ability.
  4. pink: good chewing ability.
  5. red: very good chewing ability.
Masticatory Function | Change from Baseline Change from Baseline Maximum tongue pressure status at 6-month after intervention status at 3-month after intervention
  The mixing ability was assessed using color-changeable chewing gum (Masticatory Performance Evaluating Gum XYLITOL, Lotte, Tokyo, Japan) , as follows:
  To chew as usual on the gum 120 seconds. The chewing rhythm was kept constant at once per second.color scale consisting of five intermediate colors .
  1. light green: very poor chewing ability.
  2. light yellow: poor chewing ability.
  3. light pink: no good chewing ability.
  4. pink: good chewing ability.
  5. red: very good chewing ability.
Saliva Swallowing Test(RSST) | Change from Baseline Change from Baseline Maximum tongue pressure status at 1-month after intervention
  The swallowing function states of times complete swallowing within 30 seconds was recorded using the Saliva Swallowing Test(RSST), as follows:
  participation was asked to swallow saliva as many times as possible for 30 s, while deglutition is counted through palpation of the larynx.
Saliva Swallowing Test(RSST) | Change from Baseline Change from Baseline Maximum tongue pressure status at 3-month after intervention
  The swallowing function states of times complete swallowing within 30 seconds was recorded using the Saliva Swallowing Test(RSST), as follows:
  participation was asked to swallow saliva as many times as possible for 30 s, while deglutition is counted through palpation of the larynx.
Saliva Swallowing Test(RSST) | Change from Baseline Change from Baseline Maximum tongue pressure status at 6-month after intervention
  The swallowing function states of times complete swallowing within 30 seconds was recorded using the Saliva Swallowing Test(RSST), as follows:
  participation was asked to swallow saliva as many times as possible for 30 s, while deglutition is counted through palpation of the larynx.

SECONDARY OUTCOMES:
GOHAI-T(Geriatric Oral Health Assessment Index-Taiwan) | Change from Baseline at 1 month after intervention
  The GOHAI-T of 12 questions was assessment using self-assessment oral health questionnaire.
  Have participants been totally unable to function" The scores ranged from one ("never") to five ("always"), with the total possible score ranging from 12 to 60.
GOHAI-T(Geriatric Oral Health Assessment Index-Taiwan) | Change from Baseline at 3 month after intervention
  The GOHAI-Scale of 12 questions was assessment using self-assessment oral health questionnaire.
  Have participants been totally unable to function" The scores ranged from one ("never") to five ("always"), with the total possible score ranging from 12 to 60.
GOHAI-T(Geriatric Oral Health Assessment Index-Taiwan) | Change from Baseline at 6 month after intervention
  The GOHAI-Scale of 12 questions was assessment using self-assessment oral health questionnaire.
  Have participants been totally unable to function" The scores ranged from one ("never") to five ("always"), with the total possible score ranging from 12 to 60.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Chang AH, Lin PC, Lin PC, Lin YC, Kabasawa Y, Lin CY, Huang HL. Effectiveness of Virtual Reality-Based Training on Oral Healthcare for Disabled Elderly Persons: A Randomized Controlled Trial. J Pers Med. 2022 Feb 4;12(2):218. doi: 10.3390/jpm12020218. PMID 35207706